CLINICAL TRIAL: NCT04100226
Title: Vitamin D Deficiency in Interstitial Lung Diseases
Brief Title: Vitamin D Deficiency and Effect of Its Supplementation on Interstitial Lung Diseases(ILD).
Acronym: ILD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Collaborators: Samah Selim Abdel Naiem Selim (Unknown); Naglaa Bakry Ahmed Elkhatib (Unknown)
Responsible Party: Principal Investigator, Rania Othman Ibrahim, Principle Investigator., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: N-140-2018
Record Dates: First submitted 2019-09-19; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Lung Diseases, Interstitial; Vitamin D Deficiency
Keywords: Interstitial Lung Diseases; Vitamin D Deficiency
MeSH Terms: conditions — Lung Diseases, Interstitial; Vitamin D Deficiency | interventions — Cholecalciferol; Calcium Carbonate

STUDY DESIGN:
Intervention Model Description: Arm 1(interventional group): interstitial lung diseases patients with vitamin D deficient / insufficient will receive Vitamin D supplementation and ca in addition to current treatment.
  Arm 2(control group): interstitial lung diseases patients with vitamin D deficient / insufficient will receive current treatment without vitamin D supplementation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interstitial lung patients with low vitamin D (Experimental): Arm 1:(interventional group): interstitial lung diseases patients with low vitamine D will receive Vitamin D supplementation in form of Vitamin D3 (1.25(OH)2 cholecalciferol) in dose of 200.000 IU intramuscular injection every 2 weeks for 3 months for deficient vitamin D level patients and every month for 3 months for insufficient vitamin D level patients beside ca supplementation in form ca carbonate 600 mg oral capsule once daily for 3 months for all patients in addition to current treatment.
  Interventions: Dietary Supplement: Vitamin D3 (1.25 (OH)2 cholecalciferol)
- interstitial lung diseases patients with low vitamin D (No Intervention): Arm 2(control group): interstitial lung diseases patients with vitamin D deficient / insufficient will receive their current treatment only without vitamin D supplementation.

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (1.25 (OH)2 cholecalciferol) — Vitamin D 3 in a dose of 200.000 IU intramuscular injection every 2 weeks for 3 months for Vitamin D deficient interstitial lung disease patients and every month for 3 months for vitamin D insufficient interstitial lung disease patients.
  calcium supplementation in form of ca carbonate 600 mg oral capsule once daily for 3 months for all patients.
  Other Names: calcium carbonate
  Arms: Interstitial lung patients with low vitamin D

SUMMARY:
This study evaluates serum level of Vitamin D in Interstitial Lung Diseases in patients with Interstitial Lung Diseases other than connective tissue diseases associated-Interstitial Lung Diseases and effects of its supplementation.

All patients will receive the standard regimen of treatment (corticosteroids and immunosuppressive drugs)and will be randomly assigned to either Group 1:who will receive Vitamin D supplementation (Interventional group)or Group 2:who will not receive Vitamin D supplementation(Control group).

DETAILED DESCRIPTION:
Pulmonary fibrosis was due to chronic inflammation and disordered wound healing in response to damage induced by a variety of agents such as viral infection and radiotherapy or environmental toxins.it is characterized by accumulation of myofibroblasts and excessive deposition of the extracellular matrix.Epithelial cells undergoes epithelial mesenchymal transition (EMT).

Supplementation with vitamin D or its analogs suppresses lung fibrosis via triggering anti-fibrotic effect through attenuation of transforming growth factor beta (TGF-B).vitamin D can reduce TGF-B expression and attenuate TGF-B induced epithelial mesenchymal transition in lung fibroblast and epithelial cells.

ELIGIBILITY:
Inclusion Criteria:

patients who will be diagnosed as interstitial lung disease by multidisciplinary approach based on clinical, functional, radiological and pathological diagnosis when needed.

Exclusion Criteria:

* Patients who have other diseases affecting Vitamin D levels like chronic liver diseases, chronic kidney diseases and malignancy.
* patients who will be unable to do pulmonary functions or 6-minutes walk test.
* patients with ischemic heart diseases and congestive heart failure.
* patients with connective tissue-associated interstitial lung diseases.
* interstitial lung diseases exacerbation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
change in lung functions (spirometric data) from baseline i.e change of Forced vital capacity (FVC) percent predicted values from baseline | baseline and 12 week (measurement at enrollment and end of study)
  functional improvement via improvement of pulmonary function parameters as regard to volumes like {forced vital capacity(FVC) percent predicted value} .
change in lung functions (spirometric data) from baseline i.e change of Forced expiratory volume in 1st second (FEV1) percent predicted values from baseline | baseline and 12 week (measurement at enrollment and end of study)
  functional improvement via improvement of pulmonary function parameters as regard to volumes like {forced expiratory volume in 1st second(FEV1) percent predicted value} .
change in lung functions (spirometric data) from baseline i.e change in forced expiratory flow at 25% (FEF25%) percent predicted values from baseline | baseline and 12 week (measurement at enrollment and end of study)
  functional improvement via improvement of pulmonary function parameters as regard to velocity like {forced expiratory volume in 1st second(FEV1) percent predicted value} .
change in 6-minutes walk distance | baseline and 12 week (measurement at enrollment and end of study)
  change in 6-minutes walk distance walked by the patient for 6 minutes

SECONDARY OUTCOMES:
change in dyspnea score grading from baseline | baseline and 12 week (measurement at enrollment and end of study)
  dyspnea score will be evaluated by Modified Medical Research Council(mMRC) scale which consist in 5 statements that describe almost the entire range of dyspnea from none (G 0) to almost complete in capacity ( G 4).

CONTACTS AND LOCATIONS:
Overall Officials: Esmat Ai Ali, MD, Study Chair — Professor of chest diseases,Faculty of Medicine, Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No